CLINICAL TRIAL: NCT03490708
Title: A Clinical Study of Tranilast in the Treatment of Mucinoses
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mucinoses MH Hou
Record Dates: First submitted 2018-02-04; First posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-02

CONDITIONS: Mucinoses
Keywords: Mucinoses; Tranilast
MeSH Terms: conditions — Mucinoses | interventions — tranilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tranilast (Experimental): Subjects who were treated with tranilast
  Interventions: Drug: Tranilast

INTERVENTIONS:
Drug: Tranilast — Subjects will be treated with tranilast

SUMMARY:
56 participants with Mucinoses will be selected to receive treatment of tranilast. After a period of time ,the investigators can determine the efficacy of the drug by detecting the the thickness and area of skin before and after treatment.

DETAILED DESCRIPTION:
56 participants with Mucinoses will be selected. After the signing of the informed consent ,participants will be collected the initial lesions photos,the thickness and area of skin lesions by ultrasound and magnetic resonance,and chemical examinations including blood routine examination, routine urine test, liver function, renal function. During tranilast (0.1g each time, three times a day,12 months) treatment, participants need regular follow-up (1 per month) including liver and kidney function, blood glucose level monitoring, and every three months to retest lesion thickness and area. With 3 month as a time point, participants were observed for four points. After the experiment, the experimental data will be arranged and the data of the thickness and area change of skin lesions will be statistically processed to determine whether it is meaningful.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and histopathological examination has been proved to be Mucinoses;
2. Ultrasound and magnetic resonance detection found that the skin was thickened.

Exclusion Criteria:

1. With a liver or kidney disease, or accompanied by a severe infection;
2. Poor control of primary disease;
3. With mental disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2018-04 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Measure the volume change of skin lesions by ultrasound | This experiment will last for 12 months
  During tranilast (0.1g each time, three times a day, 12 months) treatment, patients need to test lesion volume.The reduction of volume greater than 50% is judged to be effective